CLINICAL TRIAL: NCT06140186
Title: Efficacy and Safety of add-on Topical Timolol in the Management of Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor-induced Paronychia: A Prospective Randomized Open-labelled Trial
Brief Title: Efficacy and Safety of Timolol for TKI Induced Paronychia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok Wang Chun, Clinical Assistant Professor, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 23-157
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Paronychia
Keywords: EGFR TKI; Paronychia; Timolol
MeSH Terms: conditions — Paronychia | interventions — Timolol; Betamethasone Valerate

STUDY DESIGN:
Intervention Model Description: 40 Adult patients aged 18 or above who received EGFR-TKI for the treatment of NSCLC, who develop paronychia (affecting fingernails, toenails or both), will be included in this study. Patients will be randomized in 1:1 ratio using computer-generated randomization list.
Masking Description: This is an open-label trial, and no one will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Timolol combination treatment (Active Comparator): Patients will received topical timolol 0.5% eye drops (liquid form) twice daily with occlusion (i.e. covered with adhesive badge) and betamethasone valerate 0.1% cream twice daily with occlsuion for 1 month
  Interventions: Drug: Topical Timolol
- Routine arm (Active Comparator): Patients in routine arm would receive the management according to routine clinical practice, including prescription of betamethasone valerate 0.1% cream twice daily for 1 month with occlusion.
  Interventions: Drug: Betamethasone Valerate

INTERVENTIONS:
Drug: Topical Timolol — Topical timolol 0.5% eye drops (liquid form) twice daily with occlusion (i.e. covered with adhesive badge) and betamethasone valerate 0.1% cream twice daily with occlsuion for 1 month.
  Arms: Timolol combination treatment
Drug: Betamethasone Valerate — Betamethasone valerate 0.1% cream application twice daily
  Arms: Routine arm

SUMMARY:
This study would assess the clinical efficacy of add-on topical timolol 0.5% gel to betamethasone valerate 0.1% for the treatment of EGFR-TKI induced paronychia. Eligible patients, who develop paronychia (affecting fingernails, toenails or both), will be included in this study. They will be randomized in 1:1 ratio using computer-generated randomization list to receive either combination of topical timolol 0.5% gel and betamethasone valerate 0.1% lotion application twice daily or betamethasone valerate 0.1% lotion application twice daily. Patients in timolol combination treatment group will receive topical timolol 0.5% gel twice daily with occlusion (i.e. covered with adhesive badge) and betamethasone valerate 0.1% lotion twice daily with occlsuion for 1 month. Patients in routine arm would receive the management according to routine clinical practice, including prescription of betamethasone valerate 0.1% lotion twice daily for 1 month with occlusion. For patients who do not have paronychia completely resolved after 4 weeks, the treatment assigned will be continued for another 4 to 8 weeks , up to 12 weeks to see the effect.

DETAILED DESCRIPTION:
The aim of this study ist o assess the clinical efficacy of add-on topical timolol 0.5% gel to betamethasone valerate 0.1% for the treatment of EGFR-TKI induced paronychia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above, either males or females.
2. Received EGFR-TKI, namely gefitinib, erlotinib, afatinib, osimertinib, amivantamab, dacomitinib and mobocertinib.
3. Paronychia (fingernails, toenails, or both) as an adverse event from EGFR-TKI use.
4. Written informed consent obtained from patient.

Exclusion Criteria:

1. Age below18.
2. Patients who are allergic to, or contraindicated to topical timolol use.
3. Pregnant women or nursing mother.
4. Non-consenting patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
The difference in the proportion of patients achieved complete response (disappearance of the lesion, absent pain, and/or bleeding) | From baseline to month 3
  The primary outcome of this study is the proportion of patients achieved complete response (disappearance of the lesion, absent pain, and/or bleeding) on topical timolol 0.5% eye drops as compared to betamethasone valerate 0.1% cream.

SECONDARY OUTCOMES:
The proportion of patients achieved complete or partial response | From baseline to month 3
  Proportion of patients achieved complete or partial response (improvement in at least 1 of these 3 items)
Lack of response as well as proportion of patients with reduced severity of paronychia | From baseline to month 3
  Proportion of patients lack of response (improvement in less than 1 item)
Change in chronic paronychia severity index scale with treatment | From baseline to month 3
  Involvement of 1 nail fold = 1; involvement of 2 nail folds [proximal or/and lateral] = 2; bilateral lateral nail fold involvement and proximal nail fold involvement = 3), edema (absent = 0; mild = 1; moderate = 2; severe = 3), erythema (absent = 0; mild = 1; moderate = 2; severe = 3), nail plate changes (absent = 0; mild = 1; moderate = 2; severe = 3), and cuticle involvement (normal = 0; damaged = 1; absent = 2), producing a combined total score (between 0 [min.] and 14 [max.]
The improvement of paronychia by 4 point scale | From baseline to month 3
  1: 0 to <30% , 2: 30 to <50% ,3: 50 to 75% ,4: 75 to 100 % improvement)
Change in severity of pain by Visual Analog Scale | From baseline to month 3
  VAS scores ≤3.4cm corresponded to mild pain-related interference with functioning, scores of 3.5-6.4 to moderate interference, and scores ≥6.5 to severe interference.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Chun Kwok, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No